CLINICAL TRIAL: NCT05182515
Title: Interest of Plasma Exchange in Patients With Anti-interferon Type 1 Autoantibodies With Severe COVID-19 -
Brief Title: Plasma Exchange in Covid-19 Patients With Anti-interferon Autoantibodies
Acronym: EPIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20-P060
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: type 1 anti-interferon autoantibodies; Cytokine release syndrome; Plasma exchange; Pneumonia; SARS-CoV-2; Severe acute respiratory distress syndrome.
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Pneumonia; Respiratory Distress Syndrome | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: This study is an open-label, randomized, multicenter, concurrent, parallel-group, standard of care controlled, to evaluate the safety and efficacy of plasma exchange (PE) in patients with anti-interferon autoantibodies, intensive care admitted for severe or critical symptoms of respiratory illness caused by Coronavirus disease 2019 (COVID-19) defined as "Life-threatening" by the WHO scale, using a group-sequential adaptive design.
  Approximately 50 participants will be randomized 1:1 to the Investigational or Control arm. Participants randomized to the Investigational arm will receive plasma exchanges (PE) for nearly three days in addition to standard of care (SOC), while participants in the Control arm will receive SOC only. The first plasma exchange session occurs within the first 120 hours of ICU admission.
  Two interim analyses are planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care including Dexamethasone
- Therapeutic plasma exchanges (Experimental): Drug: Therapeutic plasma exchanges at day 1, 3 and 5 plus Standard of care including Dexamethasone
  Interventions: Drug: Therapeutic plasma exchange

INTERVENTIONS:
Drug: Therapeutic plasma exchange — Plasma exchange techniques reported in COVID-19 vary from study to study. No consensus exists on the use of a specific technique.
  The use of a central venous catheter will be left to the discretion of investigators. If so, central venous catheter will be inserted through the internal jugular or femoral route under ultrasound control by a trained operator. After radiographic control of the position of the catheter and the absence of complications in the placement of the catheter, plasma exchanges will be carried out.
  Three plasma exchanges of 1.5 plasma volume will be carried out every 48 hours on D1, D3 and D5. Plasma volume will be assessed by this equation VP = (1-Hct)x70xweight Body(measured). The substitution volume will be 5% albumin as first intervention. The use of a hemofiltration or centrifugation technique will be left to the discretion of each center.
  Other Names: Therapeutic plasma exchanges
  Arms: Therapeutic plasma exchanges

SUMMARY:
COVID-19 associated mortality remains high despite the advances in therapeutics such as dexamethasone. The severity of COVID-19 results from direct viral cytotoxicity, and the inflammatory response, which is associated with a hypercoagulable state, contribute to lethal hypoxemic pneumonia. During the SARS-CoV-2 replication phase, infected cells secrete chemokines and die by activating the immune system locally. A local inflammatory loop induces tissue destruction, which activates the immune system's circulating cells, leading to another amplifying loop called the cytokine storm. In these phenomena, the integrity of the interferon pathway plays a significant role.

Specific impairment of the interferon pathway has been identified in a subset of patients and is associated with high Covid-19 severity. This subset of patients presents preexisting autoimmune disease mediated by autoantibodies directed against IFN. It represents 10.2% (101/987) of patients admitted in ICU with COVID-19 pneumonia, and the observed mortality in this subgroup is 40%.

The investigators hypothesized that plasma exchanges (PE) would eliminate these autoantibodies while acting on other mechanisms of the pathogenesis of severe COVID-19, such as cytokine storm or hypercoagulability(7).

The EPIC trial aims to demonstrate the efficacy of plasma exchange in the subpopulation of patients with anti-interferon autoantibodies and severe COVID-19 hospitalized in intensive care and on oxygen therapy, high flow or not, receiving non-ventilation or invasive ventilation, on D28 survival.

DETAILED DESCRIPTION:
As of 11/09/2020, 50,000,000 people have been infected with COVID-19 worldwide, and 1,200,000 people have died, mainly from acute respiratory distress syndrome (ARDS ). Only Dexamethasone has shown survival improvement in patients hospitalized with severe COVID-19 receiving oxygen or more invasive symptomatic treatment. Despite this therapeutic advance, invasive ventilation is necessary in 30% of hospitalized cases, and mortality remains high among ventilated patients (30-40%). This study suggests that it is necessary to continue searching for a treatment to reduce this mortality rate further while confirming that immunity modulation is a promising strategy.

The severity of COVID-19 results from direct viral cytotoxicity, the accompanying inflammatory response associated with a state of hypercoagulability which contributes to lethal hypoxemic pneumonitis. During the SARS-CoV-2 replication phase, infected cells secrete chemokines and die by activating the immune system locally. A local inflammatory loop induces tissue destruction, which activates the immune system's circulating cells, leading to another amplifying loop called the cytokine storm. A high concentration of pro-inflammatory interleukins characterizes this cytokine storm. It induces an endothelial dysfunction that causes activation of the coagulation system and an increase in vascular permeability. These mechanisms lead to COVID-19 pneumopathy, and the pathologic examination reveals diffuse alveolar damage associated with a significant inflammatory infiltrate and microthrombi. These lesions cause pulmonary dysfunction and refractory hypoxia, which is the cause of mortality from COVID-19.

In these phenomena, the integrity of the type 1 interferon pathway seems to play a major role and more particularly in COVID-19. Patients in whom the type I or III interferon pathway is dysfunctional are particularly susceptible to viral damage. It is now known that dysfunction of one of the interferon pathways exposes the host to a severe viral infection such as fulminant viral hepatitis or severe influenza pneumonia caused. In a study published in September in Science, Professor Jean-Laurent Casanova's team found in 10.2% (101/987) of patients with COVID-19 pneumonia neutralizing autoantibodies directed against IFN-ω (13 patients), one of 13 types of IFN-α (36), or both (52); In this study, the authors show that these autoantibodies neutralized the ability of IFN type I to block SARS-CoV-2 infection. When a patient presents one of these autoantibodies, he is exposed to an increased mortality risk compared to the healthy population. It is estimated at 40% in the affected population versus less than 10% in the rest.

Plasma exchanges (PE) are a blood purification technique that eliminates auto-antibodies in the context of autoantibodies driven pathologies, particularly in intensive care such as autoimmune myasthenia gravis or Guillain Barré syndrome. This technique makes it possible to purify the plasma containing immunoglobulins, cytokines, chemokines, coagulation factors and replace it with plasma from healthy subjects or purified human albumin. The theoretical ability to remove some of the pro-inflammatory substances, toxins, and cellular components from the sick individual quickly identified plasma exchange as a potential therapy for COVID-19. The discovery of anti-interferon autoantibodies as a significant gravity factor leads us to hypothesize that PE would be even more beneficial in this subpopulation.

To date, eight randomized clinical trials are in progress evaluating the interest of plasma exchanges in COVID-19 on clinicaltrials.gov. The inclusion criteria in these studies are broad. As plasma exchanges are an expensive therapy with limited availability, it makes their use in all patients with severe COVID-19 impossible. In this study, the investigators propose to demonstrate the efficacy of PE in the subpopulation of patients with anti-interferon autoantibodies and severe COVID-19 hospitalized in intensive care and on oxygen therapy, high flow or not, receiving invasive or non-invasive ventilation on survival to D28.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-CoV-2 infection proven by PCR.
2. Positive detection of anti-interferon antibodies.
3. Patient, family or deferred consent (emergency clause).
4. Affiliation to a social security scheme (or exemption from affiliation). Inclusions are possible also for protected patient (under guardianship and tutornship).

Exclusion Criteria:

1. Pregnant women, parturients and nursing mothers
2. Minor patient
3. Participation in another interventional trial in progress, with the objective, even secondary, of reducing mortality
4. Indication to EPT for another associated pathology
5. Contra-indication to EPT, known allergy to albumin 5%.
6. Persons under court protection,
7. Disturbance of the haemostasis balance (PT<50%, APTT>1.5 and fibrinogen <1g/L)
8. Patient presenting a hemorrhagic diathesis (intracranial or digestive bleeding or threatening the functional prognosis)
9. Any progressive and advanced pathology whose life expectancy is less than one month
10. Bacterial or viral infectious disease (HIV) explaining most of the aggravation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-03-22 (Estimated); Study Completion 2022-03-22 (Estimated)

PRIMARY OUTCOMES:
Survival at day 28 | 28 days
  Survival up to day 28

SECONDARY OUTCOMES:
Survival at day 90 | 90 days
  Survival up to day 90
WHO Covid-19 ordinal scale at day 28 | 28 days
  Ordinal Scale for Clinical Improvement from 0 (no clinical or virological evidence of infection) to 8 (death)
WHO Covid-19 ordinal scale at day 90 | 90 days
  Ordinal Scale for Clinical Improvement from 0 (no clinical or virological evidence of infection) to 8 (death)
Lung Injury score (LIS) at day 14 | 14 days
  LIS ranges between 0 and 4, 0 points - no lung injury; 4 points severe lung injury, acute respiratory distress syndrome.
Lung Injury score at day 28 | 28 days
  LIS ranges between 0 and 4, 0 points - no lung injury; 4 points severe lung injury, acute respiratory distress syndrome.
Sequential Organ Failure Assessment day 14 | 14 days
  The SOFA Score can be used to determine the level of organ dysfunction and mortality risk in ICU patients, from 0 to 24, with severity increasing the higher the score.
Sequential Organ Failure Assessment day 28 | 28 days
  The SOFA Score can be used to determine the level of organ dysfunction and mortality risk in ICU patients, from 0 to 24, with severity increasing the higher the score.
Occurence of at least one serious adverse event | 90 days
  Grade 3 or 4 adverse events occurrence
ICU length of stay up to day 90 | 90 days
  ICU discharge date minus ICU admission date (in days)
Hospital length of stay up to day 90 | 90 days
  date of hospital discharge minus date of hospital admission
Functionnal status at day 90 according to Activities of a Daily Living score | 90 days
  The Activities of Daily Living assesses activities of daily living. A higher score indicates better activities of daily living.
Functionnal status at day 90 according to Instrumental Activities of a Daily Living score | 90 days
  The Instrumental Activities of Daily Living assesses instrumental activities of daily living. The score range is 0 to 8. A higher score indicates better instrumental activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Mazeraud Aurélien, MD, PhD, Principal Investigator — GHU Paris Psychiatrie et Neurosciences; Sharshar Tarek, MD, PhD, Study Chair — GHU Paris Psychiatrie et Neurosciences
Locations (1):
- GHU Paris Psychiatrie et Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
These documents are shared upon request to the sponsor
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, SAP and Data are shared upon request to the sponsor
Access Criteria: request to the sponsor k.sylla@ghu-paris.fr

REFERENCES:
- [Background] Tomazini BM, Maia IS, Cavalcanti AB, Berwanger O, Rosa RG, Veiga VC, Avezum A, Lopes RD, Bueno FR, Silva MVAO, Baldassare FP, Costa ELV, Moura RAB, Honorato MO, Costa AN, Damiani LP, Lisboa T, Kawano-Dourado L, Zampieri FG, Olivato GB, Righy C, Amendola CP, Roepke RML, Freitas DHM, Forte DN, Freitas FGR, Fernandes CCF, Melro LMG, Junior GFS, Morais DC, Zung S, Machado FR, Azevedo LCP; COALITION COVID-19 Brazil III Investigators. Effect of Dexamethasone on Days Alive and Ventilator-Free in Patients With Moderate or Severe Acute Respiratory Distress Syndrome and COVID-19: The CoDEX Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1307-1316. doi: 10.1001/jama.2020.17021. PMID 32876695
- [Background] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Bastard P, Rosen LB, Zhang Q, Michailidis E, Hoffmann HH, Zhang Y, Dorgham K, Philippot Q, Rosain J, Beziat V, Manry J, Shaw E, Haljasmagi L, Peterson P, Lorenzo L, Bizien L, Trouillet-Assant S, Dobbs K, de Jesus AA, Belot A, Kallaste A, Catherinot E, Tandjaoui-Lambiotte Y, Le Pen J, Kerner G, Bigio B, Seeleuthner Y, Yang R, Bolze A, Spaan AN, Delmonte OM, Abers MS, Aiuti A, Casari G, Lampasona V, Piemonti L, Ciceri F, Bilguvar K, Lifton RP, Vasse M, Smadja DM, Migaud M, Hadjadj J, Terrier B, Duffy D, Quintana-Murci L, van de Beek D, Roussel L, Vinh DC, Tangye SG, Haerynck F, Dalmau D, Martinez-Picado J, Brodin P, Nussenzweig MC, Boisson-Dupuis S, Rodriguez-Gallego C, Vogt G, Mogensen TH, Oler AJ, Gu J, Burbelo PD, Cohen JI, Biondi A, Bettini LR, D'Angio M, Bonfanti P, Rossignol P, Mayaux J, Rieux-Laucat F, Husebye ES, Fusco F, Ursini MV, Imberti L, Sottini A, Paghera S, Quiros-Roldan E, Rossi C, Castagnoli R, Montagna D, Licari A, Marseglia GL, Duval X, Ghosn J; HGID Lab; NIAID-USUHS Immune Response to COVID Group; COVID Clinicians; COVID-STORM Clinicians; Imagine COVID Group; French COVID Cohort Study Group; Milieu Interieur Consortium; CoV-Contact Cohort; Amsterdam UMC Covid-19 Biobank; COVID Human Genetic Effort; Tsang JS, Goldbach-Mansky R, Kisand K, Lionakis MS, Puel A, Zhang SY, Holland SM, Gorochov G, Jouanguy E, Rice CM, Cobat A, Notarangelo LD, Abel L, Su HC, Casanova JL. Autoantibodies against type I IFNs in patients with life-threatening COVID-19. Science. 2020 Oct 23;370(6515):eabd4585. doi: 10.1126/science.abd4585. Epub 2020 Sep 24. PMID 32972996
- [Background] Zhang Q, Bastard P, Liu Z, Le Pen J, Moncada-Velez M, Chen J, Ogishi M, Sabli IKD, Hodeib S, Korol C, Rosain J, Bilguvar K, Ye J, Bolze A, Bigio B, Yang R, Arias AA, Zhou Q, Zhang Y, Onodi F, Korniotis S, Karpf L, Philippot Q, Chbihi M, Bonnet-Madin L, Dorgham K, Smith N, Schneider WM, Razooky BS, Hoffmann HH, Michailidis E, Moens L, Han JE, Lorenzo L, Bizien L, Meade P, Neehus AL, Ugurbil AC, Corneau A, Kerner G, Zhang P, Rapaport F, Seeleuthner Y, Manry J, Masson C, Schmitt Y, Schluter A, Le Voyer T, Khan T, Li J, Fellay J, Roussel L, Shahrooei M, Alosaimi MF, Mansouri D, Al-Saud H, Al-Mulla F, Almourfi F, Al-Muhsen SZ, Alsohime F, Al Turki S, Hasanato R, van de Beek D, Biondi A, Bettini LR, D'Angio' M, Bonfanti P, Imberti L, Sottini A, Paghera S, Quiros-Roldan E, Rossi C, Oler AJ, Tompkins MF, Alba C, Vandernoot I, Goffard JC, Smits G, Migeotte I, Haerynck F, Soler-Palacin P, Martin-Nalda A, Colobran R, Morange PE, Keles S, Colkesen F, Ozcelik T, Yasar KK, Senoglu S, Karabela SN, Rodriguez-Gallego C, Novelli G, Hraiech S, Tandjaoui-Lambiotte Y, Duval X, Laouenan C; COVID-STORM Clinicians; COVID Clinicians; Imagine COVID Group; French COVID Cohort Study Group; CoV-Contact Cohort; Amsterdam UMC Covid-19 Biobank; COVID Human Genetic Effort; NIAID-USUHS/TAGC COVID Immunity Group; Snow AL, Dalgard CL, Milner JD, Vinh DC, Mogensen TH, Marr N, Spaan AN, Boisson B, Boisson-Dupuis S, Bustamante J, Puel A, Ciancanelli MJ, Meyts I, Maniatis T, Soumelis V, Amara A, Nussenzweig M, Garcia-Sastre A, Krammer F, Pujol A, Duffy D, Lifton RP, Zhang SY, Gorochov G, Beziat V, Jouanguy E, Sancho-Shimizu V, Rice CM, Abel L, Notarangelo LD, Cobat A, Su HC, Casanova JL. Inborn errors of type I IFN immunity in patients with life-threatening COVID-19. Science. 2020 Oct 23;370(6515):eabd4570. doi: 10.1126/science.abd4570. Epub 2020 Sep 24. PMID 32972995
- [Background] Hadjadj J, Yatim N, Barnabei L, Corneau A, Boussier J, Smith N, Pere H, Charbit B, Bondet V, Chenevier-Gobeaux C, Breillat P, Carlier N, Gauzit R, Morbieu C, Pene F, Marin N, Roche N, Szwebel TA, Merkling SH, Treluyer JM, Veyer D, Mouthon L, Blanc C, Tharaux PL, Rozenberg F, Fischer A, Duffy D, Rieux-Laucat F, Kerneis S, Terrier B. Impaired type I interferon activity and inflammatory responses in severe COVID-19 patients. Science. 2020 Aug 7;369(6504):718-724. doi: 10.1126/science.abc6027. Epub 2020 Jul 13. PMID 32661059
- [Background] Ciancanelli MJ, Huang SX, Luthra P, Garner H, Itan Y, Volpi S, Lafaille FG, Trouillet C, Schmolke M, Albrecht RA, Israelsson E, Lim HK, Casadio M, Hermesh T, Lorenzo L, Leung LW, Pedergnana V, Boisson B, Okada S, Picard C, Ringuier B, Troussier F, Chaussabel D, Abel L, Pellier I, Notarangelo LD, Garcia-Sastre A, Basler CF, Geissmann F, Zhang SY, Snoeck HW, Casanova JL. Infectious disease. Life-threatening influenza and impaired interferon amplification in human IRF7 deficiency. Science. 2015 Apr 24;348(6233):448-53. doi: 10.1126/science.aaa1578. Epub 2015 Mar 26. PMID 25814066
- [Background] Dupuis S, Jouanguy E, Al-Hajjar S, Fieschi C, Al-Mohsen IZ, Al-Jumaah S, Yang K, Chapgier A, Eidenschenk C, Eid P, Al Ghonaium A, Tufenkeji H, Frayha H, Al-Gazlan S, Al-Rayes H, Schreiber RD, Gresser I, Casanova JL. Impaired response to interferon-alpha/beta and lethal viral disease in human STAT1 deficiency. Nat Genet. 2003 Mar;33(3):388-91. doi: 10.1038/ng1097. Epub 2003 Feb 18. PMID 12590259
- [Background] Sancho-Shimizu V, Perez de Diego R, Jouanguy E, Zhang SY, Casanova JL. Inborn errors of anti-viral interferon immunity in humans. Curr Opin Virol. 2011 Dec;1(6):487-96. doi: 10.1016/j.coviro.2011.10.016. PMID 22347990
- [Background] Chevret S, Hughes RA, Annane D. Plasma exchange for Guillain-Barre syndrome. Cochrane Database Syst Rev. 2017 Feb 27;2(2):CD001798. doi: 10.1002/14651858.CD001798.pub3. PMID 28241090
- [Background] Gajdos P, Chevret S, Toyka K. Plasma exchange for myasthenia gravis. Cochrane Database Syst Rev. 2002;2002(4):CD002275. doi: 10.1002/14651858.CD002275. PMID 12519572
- [Background] Reeves HM, Winters JL. The mechanisms of action of plasma exchange. Br J Haematol. 2014 Feb;164(3):342-51. doi: 10.1111/bjh.12629. Epub 2013 Oct 30. PMID 24172059
- [Background] Khamis F, Al-Zakwani I, Al Hashmi S, Al Dowaiki S, Al Bahrani M, Pandak N, Al Khalili H, Memish Z. Therapeutic plasma exchange in adults with severe COVID-19 infection. Int J Infect Dis. 2020 Oct;99:214-218. doi: 10.1016/j.ijid.2020.06.064. Epub 2020 Jun 23. PMID 32585284
- [Background] Zhang L, Zhai H, Ma S, Chen J, Gao Y. Efficacy of therapeutic plasma exchange in severe COVID-19 patients. Br J Haematol. 2020 Aug;190(4):e181-e183. doi: 10.1111/bjh.16890. Epub 2020 Jun 12. No abstract available. PMID 32453903
- [Background] Lemaire A, Parquet N, Galicier L, Boutboul D, Bertinchamp R, Malphettes M, Dumas G, Mariotte E, Peraldi MN, Souppart V, Schlemmer B, Azoulay E, Canet E. Plasma exchange in the intensive care unit: Technical aspects and complications. J Clin Apher. 2017 Dec;32(6):405-412. doi: 10.1002/jca.21529. Epub 2017 Feb 1. PMID 28146331
- [Background] Tian S, Chang Z, Wang Y, Wu M, Zhang W, Zhou G, Zou X, Tian H, Xiao T, Xing J, Chen J, Han J, Ning K, Wu T. Clinical Characteristics and Reasons for Differences in Duration From Symptom Onset to Release From Quarantine Among Patients With COVID-19 in Liaocheng, China. Front Med (Lausanne). 2020 May 12;7:210. doi: 10.3389/fmed.2020.00210. eCollection 2020. PMID 32574322